CLINICAL TRIAL: NCT06658899
Title: A Phase 2, Double-Blind, Repeat-Dose, Placebo-Controlled Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CRD-4730 In Participants With Catecholaminergic Polymorphic Ventricular Tachycardia
Brief Title: A Phase 2 Study of CRD-4730 in CPVT
Acronym: CPVT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD-4730-202
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Catecholaminergic Polymorphic Ventricular Tachycardia
Keywords: CaMKII; CPVT; Ventricular Tachycardia; CRD-4730; Cardiovascular; Arrhythmia; Catecholaminergic Polymorphic Ventricular Tachycardia; CaM kinase II; Calmodulin-dependent protein kinase II
MeSH Terms: conditions — Polymorphic Catecholaminergic Ventricular Tachycardia; Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: 3-period randomized 3-sequence study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, Subject, Outcomes Assessor, and Sponsor Blinded; placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental): CRD-4730 Dose 1 Tablet
  Interventions: Drug: CRD-4730
- Dose 2 (Experimental): CRD 4730 Dose 2 Tablet
  Interventions: Drug: CRD-4730
- Dose 3 (Placebo Comparator): Placebo tablet to match CRD-4730
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRD-4730 — Oral CRD-4730 in tablet form
  Arms: Dose 1; Dose 2
Drug: Placebo — Placebo to match CRD-4730 in tablet form
  Arms: Dose 3

SUMMARY:
This is a Phase 2, multicenter, double-blind, sponsor blinded, placebo-controlled, repeat-dose clinical study of CRD-4730 to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of CRD-4730 to participants with Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT). Participants with CPVT will complete a 3-period, randomized 3-sequence study. Each participant will be randomized to one of the 3 sequences in which they will receive 2 different doses of CRD-4730 and 1 dose of matching placebo.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all the following criteria to be enrolled in this study:

1. The participant is male or female, ≥18 years of age and of legal adult age in accordance with local requirements.
2. The participant has a confirmed CPVT diagnosis, based on genetic screening for a pathogenic ryanodine receptor (RYR2) mutation and a clinical phenotype consistent with CPVT at Screening. Previous CPVT genetic testing documented in medical history is acceptable if confirmed by the Investigator and documented in the study source records.
3. The participant can perform an EST during which frequent premature ventricular contractions (PVCs; ≥10 per minute), ventricular bigeminy, or higher-grade VA (equivalent to a VA score ≥2) are identified by the Investigator.
4. The participant has been on a stable dose of at least 1 antiarrhythmic medication (including beta blockers but not amiodarone) for 4 weeks prior to Screening, unless the participant has been unable to tolerate antiarrhythmic therapy previously.
5. Adheres to all contraceptive criteria.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

1. The participant has clinically significant structural heart disease, diagnosis of heart failure, or clinically significant coronary artery disease.
2. The participant has a clinically significant abnormal ECG not explained by the diagnosis of CPVT at Screening or clinically significant abnormal intervals, such as prolonged QT.
3. The participant has a history of a myocardial infarction, cerebrovascular accident, or transient ischemic attack within 3 months of Screening.
4. The participant undergoes implantable cardioverter-defibrillator (ICD) implantation or has sympathetic nerve denervation within 3 months of Screening.
5. The participant has an anticipated change in exercise regimen or new exercise program during the course of the study.
6. The participant has a history of malignancy within the past 5 years at Screening, with the exception of successfully treated basal cell carcinoma or nonmetastatic squamous cell carcinoma of the skin or cervical carcinoma in situ. Prior exposure to chest radiation for any malignancy is exclusionary.
7. The participant has abnormal blood pressure, defined as supine symptomatic hypotension, systolic blood pressure >150 mm Hg or diastolic blood pressure >90 mm Hg, or symptomatic bradycardia or a heart rate >100 bpm at Screening and/or on Day 1. Blood pressure and pulse should be measured after the participant has been in the seated position after 5 minutes of rest.
8. The participant has hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × (upper limit of normal [ULN]) and/or total bilirubin >1.5 × ULN at Screening (unless secondary to confirmed Gilbert syndrome).
9. The participant has acute or chronic hepatitis B (HBV; defined as hepatitis B surface antigen [HBsAg] reactive), acute or chronic hepatitis C virus (HCV; defined as detection of HCV antibody and RNA [qualitative]), or human immunodeficiency virus (HIV) infection.
10. The female participant is pregnant, lactating/breastfeeding, or has plans to become pregnant during the study or within 3 months following the last study drug administration.
11. The participant has taken any antiarrhythmic drug in addition to their stable, chronic regimen unless it has been at least 5 half-lives since administration at the time of Screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures | Baseline to Day 101
  The number and severity of treatment-emergent adverse events (TEAEs) related to study drug treatment

SECONDARY OUTCOMES:
Secondary Outcome Measure | Baseline to Day 15; Baseline to Day 44; Baseline to Day 73
  Change in VA score during EST from baseline to Day 15, from baseline to Day 44, and from baseline to Day 73
Secondary Outcome Measures | Baseline to Day 15; Baseline to Day 44; Baseline to Day 73
  Plasma concentrations of CRD-4730 over time for each treatment period

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Cardurion Investigative Site, San Francisco, California
  - Cardurion Investigative Site, Morrisville, North Carolina
  - Cardurion Investigative Site, Houston, Texas
  - Cardurion Investigative Site, Madison, Wisconsin
- Cardurion Investigative Site, Saint-Herblain, France
- Cardurion Investigative Site, Pavia, Pavia, Italy
- Cardurion Investigative Site, Amsterdam, North Holland, Netherlands
- Cardurion Investigative Site, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takagahara, Shuichi, et al. "Novel, Potent, and Highly Selective Calcium/Calmodulin-Dependent Protein Kinase II (CaMKII) Inhibitors Reduce Substrate Phosphorylation in Rat Hearts and Prolong Survival in a Mouse Model of Severe Heart Failure." Circulation 148.Suppl_1 (2023): A12726-A12726.